CLINICAL TRIAL: NCT05635331
Title: Early Treatment of Heart Failure: a Non-interventional Observational Study Program of Patients With Heart Failure and Initiated on Dapagliflozin (EVOLUTION-HF - GREECE)
Brief Title: Real-world Dapagliflozin Experience in Patients With Heart Failure in Greece
Acronym: EVOLUTION-HF
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1699R00046
Record Dates: First submitted 2022-11-23; First posted 2022-12-02 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

SUMMARY:
Heart failure (HF) is a global, public health issue that affects more than 63 million people worldwide. Despite advancements in treatment, a HF diagnosis still leads to significant morbidity and mortality. Dapagliflozin has been approved by both the US Food and Drug Administration (FDA) and the European Medicines Agency (EMA), in May 2020 and November 2020 respectively, for HF with reduced ejection fraction (HFrEF). The overall aim of this study is to describe the characteristics of patients initiating dapagliflozin for the treatment of HFrEF and to provide early insights into real-world dapagliflozin treatment patterns as well as patient-reported outcomes (PROs) including quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years as of study index date; the study index date is the date of initiation of treatment with dapagliflozin
* Patient received/receiving treatment with dapagliflozin for Heart Failure with reduced Ejection Fraction in accordance with the local dapagliflozin product label
* Signed and dated informed consent prior to enrolment in the study

Exclusion Criteria:

* Patient is enrolled less than 14 days or more than 60 days following initiation of dapagliflozin
* Prior treatment with dapagliflozin or other Sodium Glucose co-transporter 2 inhibitor treatment
* Initiation of dapagliflozin outside of local Heart Failure label
* Diagnosis of Type 1 diabetes prior to enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have received treatment with dapagliflozin for Heart Failure with reduced Ejection Fraction will be eligible for enrolment by physicians from outpatient and inpatient settings. Eligible patients will be selected after they have been identified in paper or electronic medical records by the participating investigator. Consecutive patients prescribed dapagliflozin should be identified by the investigator and, unless failing to meet the inclusion and exclusion criteria, should be invited to participate. Patients will only be enrolled after they have given consent to participate in the study.
  In all cases, the decision to treat a patient with dapagliflozin must be made prior to the decision to enroll the patient into the study. To help ensure this, at least 14 days must have elapsed (but no more than 60 days) from the date of initiation of dapagliflozin before a patient can be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2022-12-28 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Baseline characteristics (demographic and clinical) | Baseline to 12 months
  To describe the baseline demographic and clinical characteristics of patients newly prescribed dapagliflozin for the treatment of Heart Failure with reduced Ejection Fraction
Time to discontinuation of dapagliflozin | Baseline to 12 months
  Time from dapagliflozin treatment initiation until the time at which participants stop taking the medication for any reason.
Number of reasons for dapagliflozin treatment discontinuation | Baseline to 12 months
  Number of reasons for dapagliflozin treatment discontinuation as noted by a health care professional will be extracted and described as the number and proportion of participants who have discontinued dapagliflozin according to each reasons presented.
Number of dapagliflozin treatment changes | Baseline to 12 months
  The number of participants who switch from dapagliflozin to another Heart Failure medication.
Time to other HF medication discontinuation | Baseline 12 months
  Time from initiation of heart failure medication other than dapagliflozin until the time at which participants discontinued treatment with that medication.
Number of other heart failure treatment dosage changes | Baseline to 12 months
  The number of participants with dosage changes for heart failure medication other than dapagliflozin.
Number of other heart failure treatment initiation | Baseline to 12 months
  The number of participants who initiate new heart failure medication other than dapagliflozin.

SECONDARY OUTCOMES:
Absolute change from baseline in Kansas City Cardiomyopathy Questionnaire (KCCQ) score | Measured at enrollment and 3, 6, 9 and 12 months
  The KCCQ is a 23-item questionnaire that quantifies physical limitations, self-efficacy, social interference and quality of life. Summary scores will be examined at each assessment point during follow-up. For each of the assessment periods, descriptive statistics for the observed value, change from baseline and the 95% two-sided confidence interval for the mean change will be presented. The proportions of participants with overall health status classified as poor, fair, good, and excellent will be examined at each assessment point. Additionally, the proportions of participants who experience clinically meaningful changes in overall health status: improvement (≥5 point increase), deterioration (≥5 point decrease), and stable (<5 point increase or decrease) will be examined at each assessment point.
Absolute change from baseline in Medication Adherence Report Scale (MARS)-5 questionnaire | Measured at enrollment, 3, 6, 9 and 12 months
  The MARS-5 is five-item self-report adherence scale which assesses both intentional and non-intentional non-adherence. Respondents rate the frequency with which the five different medication-taking behaviors occur, scoring each item on a 1-5-point scale with higher scores indicating higher reported adherence.

CONTACTS AND LOCATIONS:
Locations (7):
- Greece (7):
  - Research Site, Alexandroupoli
  - Research Site, Athens
  - Research Site, Chania
  - Research Site, Heraklion
  - Research Site, Ioannina
  - Research Site, Pátrai
  - Research Site, Thessaloniki

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1699R00046&attachmentIdentifier=27b8a2eb-3a54-499d-a4c8-5a95abec7701&fileName=D1699R00046_Redacted_CSR_Synopsis.pdf&versionIdentifier=